CLINICAL TRIAL: NCT01612897
Title: Computer Assisted Autism Care (CAAC)
Brief Title: Study of the Effectiveness of a Computer Decision Support System to Improve Physicians' Screening for Autism
Acronym: CAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: R01HS018453 (AHRQ)
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Children Undergoing Routine Care; Children With Autism
Keywords: autism; well child care; screening; computer; reminders
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer based reminders to MD (Experimental): Children in this arm attend a clinic that is randomly assigned to receive physician alerts to screen appropriate children for autism.
  Interventions: Other: Computer based care reminders
- Usual care arm (No Intervention): Children in this are receive usual care from a clinic randomly chosen to serve as a control.

INTERVENTIONS:
Other: Computer based care reminders — Physicians in the intervention clinic will receive computer generated reminders to screen for autism among children of appropriate age visiting the clinic.
  Arms: Computer based reminders to MD

SUMMARY:
The investigators hypothesize that children seen in a clinic that uses a compute based system known as CHICA, which reminds pediatricians to screen at defined time point for autism, will be screened more consistently for autism and receive more timely diagnostic a treatment services.

DETAILED DESCRIPTION:
To be eligible for this trial, participants must receive their care at one of four primary care clinics in Indianapolis where the CHICA system is used.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy children receiving routine care in one of four clinics in Indianapolis who participate in this study.

Exclusion Criteria:

* Previously known autism spectrum disorders or other causes of developmental delay

Ages: 17 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 368 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Structure autism screening instrument administered | Up to 4 years
  Physicians are reminded by the computer system to screen children under 3 years of age for autism with a structured screening instrument. Chart abstraction is used to document whether or not the screening occurred.

SECONDARY OUTCOMES:
Are appropriate diagnostic studies conducted among children who screen positive for autism. | Up to 4 years
  Among children who a suspected of having autism, chart abstraction and interviews are done to determine if the child received appropriate diagnostic and studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Wishard (Eskenazi) Healthcare clinics, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Downs SM, Bauer NS, Saha C, Ofner S, Carroll AE. Effect of a Computer-Based Decision Support Intervention on Autism Spectrum Disorder Screening in Pediatric Primary Care Clinics: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1917676. doi: 10.1001/jamanetworkopen.2019.17676. PMID 31851348